CLINICAL TRIAL: NCT03067792
Title: FOLFIRI Versus Docetaxel and Cisplatin as a Second-line Chemotherapy After Failure of First-line Chemotherapy in Advanced Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 4-2014-0626
Record Dates: First submitted 2017-02-22; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Inoperable Gastric Cancer
Keywords: inoperable gastric cancer; palliative chemotherapy
MeSH Terms: interventions — Fluorouracil; Irinotecan; Leucovorin; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFIRI (Active Comparator): 2nd palliative chemotherapy with FOLFIRI regimen,In FOLFIRI group, patients received irinotecan 180 mg/m2 and 5- fluorouracil 400mg/m2 intravenously bolus injection on days 1 and leucovorin 200mg/m2 for 2 hours and 5-fluorouracil 600mg/m2 for 22 hours intravenously infusion on day 2 of a 14-day cycle. Response evaluation would be done after 3 cycle of chemotherapy in DP group
  Interventions: Drug: 5-fluorouracil, irinotecan and leucovorin
- DP (Active Comparator): 2nd palliative chemotherapy with Docetaxel/cisplatin regimen, In DP group, patients received docetaxel 75 mg/m2 and cisplatin 75mg/m2 intravenously on days 1 of a 21-day cycle. Response evaluation would be done after 2 cycle of chemotherapy in DP group
  Interventions: Drug: docetaxel and cisplatin

INTERVENTIONS:
Drug: 5-fluorouracil, irinotecan and leucovorin — In FOLFIRI group, patients received irinotecan 180 mg/m2 and 5-fluorouracil 400mg/m2 intravenously bolus injection on days 1 and leucovorin 200mg/m2 for 2 hours and 5-fluorouracil 600mg/m2 for 22 hours intravenously infusion on day 2 of a 14-day cycle.
  Arms: FOLFIRI
Drug: docetaxel and cisplatin — In DP group, patients received docetaxel 75 mg/m2 and cisplatin 75mg/m2 intravenously on days 1 of a 21-day cycle.
  Arms: DP

SUMMARY:
Patients diagnosis with inoperable gastric cancers are treated with palliative chemotherapy.

Palliative chemotherapy had proven to be better overall survivals and quality of life in unresectable advanced gastric cancer. NCCN guideline suggested two or three drug cytotoxic regimen as a first line therapy. But response rate of those regimens is about 50 percent. Disappointingly most of cases are about to experience progression of disease.

Second line regimens of palliative chemotherapy are also have shown its efficacy and recommended within patients with better performance status. But There is still lack of evidences in gastric cancer patients second line chemotherapy. Several phase II trial those subjects are 2nd line palliative chemotherapy in gastric cancer had suggested that irinotecan, taxane, oxaliplatin, oral fluorouracil.Investigator assessed whether cisplatin in combination with paclitaxel would increase response rate in patient previously treated for advanced gastric cancer compared with FOFIRI regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 19 years old and younger than 75 years old
2. Pathologically confirmed gastric cancer
3. Inoperable stage at diagnosis
4. experienced diseases progression in first line palliative chemotherapy
5. ECOG performance status 0 or 1
6. Adequate renal function (serum creatinine < 1.5 mg/dL or calculated creatinine clearance ≥ 60 ml/min)
7. Adequate liver function (total bilirubin < 1.5 X the upper limits of normal (ULN), AST and ALT <3 X UNL, and alkaline phosphatases < 3 X ULN or < 5 x ULN in case of liver involvement)
8. Adequate BM function (WBC ≥ 3,500/µl, absolute neutrophil cell count ≥ 1,500 /µl, platelet count ≥ 100,000/µl)
9. Subjects who given written informed consent after being given a full description of the study

Exclusion Criteria:

1. double primary cancer other than gastric cancer
2. history of palliative radiation therapy
3. Pregnant or on breast feeding
4. Neuropathy grade > 3
5. Active infection
6. Symptomatic cardiopulmonary diseases
7. Active hepatitis of liver cirrhosis
8. Impaired renal function
9. Impaired psychologic bone marrow function
10. Psychologic disorder, Severe neurologic disorder.
11. hypersensitivity to chemotherapeutic agent

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2016-10-17 (Actual)

PRIMARY OUTCOMES:
response rate | up to 2 year
  CT examination would be done at 7~8 weeks after initiation of 1st cycle chemotherapeutic agent, After 2 cycle of chemotherapy in DP group and 3cyle of chemotherapy in FOFIRI group.

SECONDARY OUTCOMES:
diseases control rate | up to 2 year
  disease control, defined as the proportion of patients who had a best response of complete response, partial response, or stable
Overall survival | up to 2 year
  overall survival, defined as time from randomisation to death
progression free survival | up to 2 year
  progression-free survival, defined as time from randomisation to radiographic progression or death

IPD SHARING:
Plan to Share IPD: No